CLINICAL TRIAL: NCT05261724
Title: Contribution of Diffusion Tensor Imaging and Tractography in Primary and Secondary Brain Tumors Evaluation
Brief Title: Diffusion-tensor Imaging in Brain Tumors Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other)
Responsible Party: Principal Investigator, Mihail Porutiu, Phd student, George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures
Other Study IDs: GEPaladeU
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Diffusion Tensor Imaging; Tractography; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary brain tumors
  Interventions: Diagnostic Test: MRI
- Patients with secondary brain tumors
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — In this study patients with suspected primary and secondary brain tumors, confirmed by routine MRI evaluation (T1, T2, T2*, FLAIR, T1 with contrast sequences) will undergo DWI and DTI evaluation.

SUMMARY:
Primary and secondary brain tumors are challenging pathologies regarding diagnosis and treatment. MRI is widely used in the imaging evaluation and surgical planning, due to its spatial resolution and ability of tissular characterization.

In this study patients with suspected brain tumors, confirmed by routine MRI evaluation (T1, T2, T2*, FLAIR, T1 with contrast sequences) will undergo DWI and DTI evaluation. By analyzing collected data from MRI evaluation and patient records regarding surgical and histopathological data our aim is to investigate derived imaging biomarkers with impact in the surgical planning and rehabilitation of the patients.

ELIGIBILITY:
Inclusion Criteria:

* brain tumors confirmed by routine MRI evaluation
* surgical treatment with histopathological diagnosis

Exclusion Criteria:

* MRI contraindications
* past or present neurological or neurosurgical condition, beside the tumor
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected primary or secondary brain tumors, confirmed by routine MRI evaluation followed by surgical treatment and histopathological exam.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2022-03-14 (Estimated)

PRIMARY OUTCOMES:
Tract damage | 3 months
  Assess the damage of tracts at baseline preoperative

SECONDARY OUTCOMES:
Craniotomy size | 3 months
  Assess the size of craniotomy in patients with postoperative CT follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Porutiu, Principal Investigator — George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures
Locations (1):
- SCJU Mures, Târgu Mureş, Mureș County, Romania